CLINICAL TRIAL: NCT06019000
Title: A Randomized, Double-Blinded, Placebo-Controlled Trial to Determine The Safety and Efficacy of CYR-064
Brief Title: Study of CYR-064 Versus Placebo in Patients.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cyrano Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYR-064-01
Record Dates: First submitted 2023-05-11; First posted 2023-08-31 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Hyposmia
Keywords: post viral smell loss
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Intervention Model Description: The study treatment of CYR-064 is administered for a 24-week Treatment Period. Patients who meet all study criteria and have consented to participation will be randomized (1:1:1) to three parallel study arms, with two different dose strengths and a placebo group over 24 weeks.
  CYR-064 dose 1 CYR-064 dose 2 Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There will be a placebo match and blinded randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- CYR-064 dose 1 (Active Comparator): Treatment with nasal solution of CYR-064 twice a day for 24 weeks. CYR-064 will be self-administered by patients.
  Interventions: Combination Product: CYR-064
- CYR-064 dose 2 (Experimental): Treatment with nasal solution of CYR-064 twice a day for 24 weeks. CYR-064 will be self-administered by patients.
  Interventions: Combination Product: CYR-064
- Placebo (Placebo Comparator): Treatment with Placebo nasal solution for 24 weeks. CYR-064 will be self-administered by patients.
  Interventions: Combination Product: CYR-064

INTERVENTIONS:
Combination Product: CYR-064 — CYR-064 is a nasal solution.

SUMMARY:
Randomized, double-blinded, placebo-controlled trial to determine the safety and efficacy of CYR-064.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and effectiveness of CYR-064 in a randomized, double-blinded, placebo-controlled trial to determine the safety and efficacy of CYR064.

The study will take approximately 32 weeks which will include a 4-week screening period to evaluate if participants are right for the Study, followed by a 24-week Treatment Period, and a 1 week follow up after participants have completed the Study. About 150 subjects will participate in this study in about 25 research sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent.
* Male or female 18-70 years of age.
* Endoscopy of the nasal cavity showing no structural or pathologic issues leading to hyposmia (nasal polyps, sinusitis, infection, etc.) that in the opinion of the Investigator, believes would hinder the delivery of study drug to the olfactory receptors.
* CT scan of the nasal cavity after the onset of hyposmia (within prior 2 years) prior to Baseline showing no structural or pathologic issue leading to hyposmia that in the opinion of the Investigator, believes would hinder the delivery of study drug to the olfactory receptors.
* Willing and able to self-administer the study drug, follow the study drug administration instructions, comply with study procedures, and participate in the scheduled study visits specified in this protocol.

Exclusion Criteria:

* History of traumatic brain injury, Parkinson's disease, early dementia, Alzheimer's disease, or any other condition in which hyposmia is not expected to improve in the opinion of the Investigator, such as history of congenital or idiopathic hyposmia or a surgical procedure that led to hyposmia.
* History of surgery that led to hyposmia.
* Concomitant Medical Conditions
* Current symptoms or signs of an acute respiratory viral illness at Screening or Baseline.
* Chronic viral infection or immunodeficiency condition (e.g., medical history of human immunodeficiency virus) based on medical records.
* Any active malignancy.
* Any concomitant medical condition that in the opinion of the Investigator, compromises patient safety or compliance with the study protocol or collected data.
* History of moderate to severe Substance Use Disorder within the past 3 years as assessed by the Investigator.
* History of persistent chronic sinusitis without polyps or chronic sinusitis with polyps.
* Use or planned use of tobacco or nicotine-containing products, including smoking, smokeless tobacco, e-cigarettes, or nicotine replacement products within 3 months prior to Screening through EOS.
* Unwilling or unable to discontinue current or planned use of over the counter or prescription medication administered intranasally, with the exception of nasal saline.
* Use or planned use of another investigational drug within 4 weeks prior to Screening through Follow-Up.
* Receiving any concomitant medication/therapy that would, in the opinion of the Investigator, compromise patient safety or compliance with the study protocol or collected data.
* General Exclusions Any female who is pregnant, planning to become pregnant during the study, or who is lactating.

Vulnerable patients. Any condition or abnormality (including clinical laboratory, physical examination, or vital sign abnormalities), current or past, that, in the opinion of the Investigator, would compromise the efficacy evaluation, safety of the patient, or would interfere with or complicate study procedures or assessments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome - Safety and Tolerability | Approximately 32 weeks
  The count and percentage of patients reporting AEs, SAEs, and SUSARs will be summarized overall, by System Organ Class, Preferred Term within the System Organ Class, maximum severity, and relationship to study drug. All other safety parameters, including clinical laboratory values through blood draws, will be summarized using descriptive statistics for continuous variables and counts and percentages for categorical variables. All changes in nasal mucosal appearance will be noted.

SECONDARY OUTCOMES:
Secondary Outcome-improvement on NRS-11 Smell-PRO | Approximately 24 weeks
  Improvement in patient reported NRS-11 Smell-PRO (scale of 0-10) in CYR-064 low dose and high dose groups as compared with placebo from Baseline to Week 24.
Secondary Outcome-improvement on NRS-11 Taste-PRO | Approximately 24 weeks
  Improvement in patient reported NRS-11 Taste-PRO (scale of 0-10) in CYR-064 low dose and high dose groups as compared with placebo from Baseline to Week 24.
Secondary Outcome-Mean Change in NRS-11 Smell-PRO | Approximately 24 weeks
  Mean Change in NRS-11 Smell-PRO from Baseline to Week 24 between CYR-064 low and high dose and placebo from Baseline to Week 24
Secondary Outcome-Mean Change in NRS-11 Taste-PRO | Approximately 24 weeks
  Mean Change in NRS-11 Taste-PRO from Baseline to Week 24 between CYR-064 low and high dose and placebo from Baseline to Week 2
Change in Visual Rating Scale (VRS) scores | Approximately 24 weeks
  Change in Visual Rating Scale (VRS) scores in CYR-064 low dose and high dose groups as compared with placebo from Baseline to Week 24.
  * VRS high dose versus placebo
  * VRS low dose versus placebo
  * VRS low and high dose combined versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Mas Takashima, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (14):
- United States (14):
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - ENTAAFL, Boca Raton, Florida
  - ENTAAFL, Plantation, Florida
  - ENTAAFL, Port Saint Lucie, Florida
  - Rush University Medical Center, Chicago, Illinois
  - KU Medical Center-University of Kansas, Kansas City, Kansas
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Tandem Clinical Research, Marrero, Louisiana
  - Centers for Advanced ENT, Baltimore, Maryland
  - Specialty Physician Associates, Bethlehem, Pennsylvania
  - Medical University of South Carolina-MUSC, Charleston, South Carolina
  - Charleston ENT and Allergy, North Charleston, South Carolina
  - Houston Methodist, Houston, Texas
  - Ear Nose Throat & Allergy Associates, Puyallup, Washington

IPD SHARING:
Plan to Share IPD: No
Descriptive statistics

REFERENCES:
- [Background] Henkin RI, Levy LM, Fordyce A. Taste and smell function in chronic disease: a review of clinical and biochemical evaluations of taste and smell dysfunction in over 5000 patients at The Taste and Smell Clinic in Washington, DC. Am J Otolaryngol. 2013 Sep-Oct;34(5):477-89. doi: 10.1016/j.amjoto.2013.04.006. Epub 2013 Jun 2. PMID 23731850
- [Background] Henkin RI. Comparative monitoring of oral theophylline treatment in blood serum, saliva, and nasal mucus. Ther Drug Monit. 2012 Apr;34(2):217-21. doi: 10.1097/FTD.0b013e3182492a20. PMID 22377744
- [Background] Henkin RI. Growth Factors in Olfaction. In: Preedy VR, editor. Handbook of Growth and Growth Monitoring in Health and Disease. New York, NY: Springer New York; 2012. p. 1417-36.
- [Background] Henkin RI, Abdelmeguid M. Improved Smell and Taste Dysfunction with Intranasal Theophylline. Am J Otolaryngol Head Neck Surg. 2019;2(9):1070.
- [Background] Henkin RI, Hosein S, Stateman WA, Knoppel AB, Abdelmeguid M. Improved smell function with increased nasal mucus sonic hedgehog in hyposmic patients after treatment with oral theophylline. Am J Otolaryngol. 2017 Mar-Apr;38(2):143-147. doi: 10.1016/j.amjoto.2016.11.010. Epub 2016 Nov 23. PMID 27923495
- [Background] Henkin RI, Schultz M, Minnick-Poppe L. Intranasal theophylline treatment of hyposmia and hypogeusia: a pilot study. Arch Otolaryngol Head Neck Surg. 2012 Nov;138(11):1064-70. doi: 10.1001/2013.jamaoto.342. PMID 23165381
- [Background] Henkin RI, Velicu I. cAMP and cGMP in nasal mucus related to severity of smell loss in patients with smell dysfunction. Clin Invest Med. 2008;31(2):E78-84. doi: 10.25011/cim.v31i2.3367. PMID 18377764
- [Background] Henkin RI, Velicu I, Schmidt L. An open-label controlled trial of theophylline for treatment of patients with hyposmia. Am J Med Sci. 2009 Jun;337(6):396-406. doi: 10.1097/MAJ.0b013e3181914a97. PMID 19359985
- [Background] Henkin RI, Velicu I, Schmidt L. Relative resistance to oral theophylline treatment in patients with hyposmia manifested by decreased secretion of nasal mucus cyclic nucleotides. Am J Med Sci. 2011 Jan;341(1):17-22. doi: 10.1097/MAJ.0b013e3181f1fdc8. PMID 21191261